CLINICAL TRIAL: NCT00451139
Title: Ototoxicity of Artemether / Lumefantrine (Coartem) and Other Antimalarials
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Jimma University (Other)
Collaborators: Ludwig-Maximilians - University of Munich (Other)
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: AITM0107
Record Dates: First submitted 2007-03-21; First posted 2007-03-23 (Estimated); Last update posted 2007-03-23 (Estimated); Status verified 2007-03

CONDITIONS: Malaria
MeSH Terms: conditions — Malaria | interventions — Artemether, Lumefantrine Drug Combination; Quinine; atovaquone, proguanil drug combination

INTERVENTIONS:
Drug: artemether/lumefantrine
Drug: quinine
Drug: atovaquone/proguanil

SUMMARY:
The purpose of the study is to evaluate the potential side-effects of artemether / lumefantrine and other antimalarials on the auditory function.

DETAILED DESCRIPTION:
Artemisinin based combination therapies (ACT) currently are the most promising treatment options for uncomplicated falciparum malaria. There have been controversial reports about possible ototoxicity of artemether / lumefantrine (Coartem®) from retrospective studies. In this investigation treatment of uncomplicated malaria with artemether / lumefantrine, quinine, where side-effects on hearing are known, or atovaquone / proguanil, where no such effects have been reported, are compared. Auditoy function is examined (Auditory Brainstem Response, Pure-tone Audiometry, Otoacustic Emissions) before treatment, after 7, 28, and, for determination of irreversibility, after 90 days.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged above 5 years
* Uncomplicated falciparum malaria
* Axillary Temperature ≥37,5°C or history of fever within the previous 24 hours
* Ability to tolerate oral therapy
* Informed consent by the patient or by parent/guardian for children
* Residence in study area

Exclusion Criteria:

* Known or suspected hearing deficits
* Adequate anti-malarial treatment within the previous 7 days
* Mixed infection
* Danger signs and signs of severe malaria as defined by the WHO
* Presence of severe underlying disease (cardiac, renal, hepatic diseases, malnutrition, known HIV infection)
* Concomitant disease masking assessment of response
* History of allergy or intolerance against study medications
* Pregnancy

Min Age: 5 Years | Sex: All
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Nebreed Fesseaha, MD, Dean, Study Chair — Facuty of Medical Sciences Jimma University
Locations (1):
- Jimma University Hospital, Jimma, Ethiopia